CLINICAL TRIAL: NCT04931862
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 1b/2a Study of WVE-004 Administered Intrathecally to Patients With C9orf72-associated Amyotrophic Lateral Sclerosis (ALS) or Frontotemporal Dementia (FTD)
Brief Title: Study of WVE-004 in Patients With C9orf72-associated Amyotrophic Lateral Sclerosis (ALS) or Frontotemporal Dementia (FTD)
Acronym: FOCUS-C9
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Despite robust, sustained reductions in poly(GP), no clinical benefit was seen at 24 weeks, and reductions in poly(GP) were not associated with stabilization in functional outcomes. Based on these data, Wave decided to stop development of WVE-004.
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-004-001
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: ALS; FTD

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- WVE-004 (Dose A) or placebo (Experimental)
  Interventions: Drug: WVE-004; Drug: Placebo
- WVE-004 (Dose B) or placebo (Experimental)
  Interventions: Drug: WVE-004; Drug: Placebo
- WVE-004 (Dose C) or placebo (Experimental)
  Interventions: Drug: WVE-004; Drug: Placebo
- WVE-004 (Dose D) or placebo (Experimental)
  Interventions: Drug: WVE-004; Drug: Placebo

INTERVENTIONS:
Drug: WVE-004 — WVE-004 is a stereopure antisense oligonucleotide (ASO)
Drug: Placebo — Artificial cerebrospinal fluid (aCSF)

SUMMARY:
This is a Phase 1b/2a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and PD of intrathecal (IT) WVE-004 in adult patients with C9orf72-associated ALS or FTD. To participate in the study, patients must have a documented mutation (GGGGCC [G4C2] repeat expansion) in the first intronic region of the C9orf72 gene and be diagnosed with ALS or FTD.

ELIGIBILITY:
Inclusion Criteria:

1. ALS-specific: Diagnosis of ALS based on clinical manifestations.
2. ALS-specific: Clinically diagnosed possible, laboratory supported probable, probable, or definite criteria for diagnosing ALS according to the World Federation of Neurology revised El Escorial criteria.
3. ALS-specific: Patients receiving riluzole have been on a stable dose for a minimum of 30 days.
4. ALS-specific: Patients on edaravone have received a minimum of 1 cycle (28 days).
5. ALS-specific: Patients discontinuing riluzole or edaravone had the last dose administered ≥1 month prior to Screening.
6. FTD-specific: Must have Global Clinical Dementia Rating - Frontotemporal Lobar Degeneration (CDR® plus NACC FTLD) score of 0.5 or 1.
7. FTD-specific: Able to undergo periodic magnetic resonance imaging (MRI) of the brain. Participants with mixed phenotype (ALS and FTD) need not undergo MRI if their ALS symptoms prevent it.
8. Mixed-phenotype: Patients who are mixed phenotype (ALS and FTD) must meet both the ALS-specific and FTD-specific criteria.

Exclusion Criteria:

1. Clinically significant medical finding on the physical examination other than C9orf72-associated ALS or FTD that, in the judgment of the Investigator, will make the patient unsuitable for participation in, and/or completion of the trial procedures
2. Received any other investigational drug, biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Received an investigational oligonucleotide, within the past 6 months or 5 half-lives of the drug, whichever is longer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Safety: Proportion of patients with adverse events (AEs) | Period 1 Day 1 to Period 2 Week 24 (end of study)

SECONDARY OUTCOMES:
Pharmacokinetic: Concentration of WVE-004 in cerebrospinal fluid (CSF) | Period 1 Day 1 to Period 2 Week 24 (end of study)
Pharmacodynamic: Change from baseline in concentration of poly-GP levels in the CSF | Period 1 Day 1 to Period 2 Week 24 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (17):
- Australia (3):
  - Macquarie University, North Ryde, New South Wales
  - The Wesley Hospital, Brisbane, Queensland
  - Perron Institute, Nedlands, Western Australia
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Center - Research Institute, Montreal, Quebec
- St James Hospital - Ireland, Dublin, Ireland
- Netherlands (2):
  - Erasmus University MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - New Zealand Brain Research Institute, Christchurch
- Karolinska University Hospital, Solna, Sweden
- United Kingdom (5):
  - University of Cambridge, Cambridge
  - University College London Hospital, London
  - King's College Hospital, London
  - University of Oxford - Nuffield Department of Clinical Neurosciences, Oxford
  - University of Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: No